CLINICAL TRIAL: NCT00834392
Title: A Pilot Study of Exercise in Men With Prostate Cancer Receiving Androgen Depletion Therapy
Brief Title: Exercise in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: C. Ellen Lee, PhD, PT, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2008:035
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Walking exercise
  Arms: Exercise

SUMMARY:
The purpose of this pilot study is to compare a walking exercise program (Exercise Group) to standard medical care (Control Group) in prostate cancer survivors receiving androgen depletion therapy (ADT). The central hypothesis of the proposed research is that the walking exercise program will have a positive impact on the bone health, health-related quality of life, and physical function of men with prostate cancer receiving ADT.

ELIGIBILITY:
Inclusion Criteria:

* men aged 50 years or older
* diagnosed with adenocarcinoma prostate cancer
* will initiate and receive continuous ADT (luteinizing hormone releasing hormone agonist (LHRH) or combination of LHRH and anti-androgen) for at least 12 months after recruitment
* Patients will also consent to participating in the study.

Exclusion Criteria:

* severe cardiac disease (New York Heart Association class III or greater)
* angina
* severe osteoporosis
* uncontrolled hypertension (blood pressure > 160/95mm Hg)
* orthostatic blood pressure drop > 20mm Hg
* moderate to severe aortic stenosis
* acute illness or fever
* uncontrolled atrial or ventricular dysrhythmias
* uncontrolled sinus tachycardia (> 120 beats per minute)
* uncontrolled congestive heart failure third-degree atrio-ventricular heart block, active pericarditis or myocarditis, recent embolism, thrombophlebitis, deep vein thrombosis, resting ST displacement (> 3mm), uncontrolled diabetes, uncontrolled pain, cognitive impairment, history of falls due to balance impairment or lost of consciousness, severe neuromusculoskeletal conditions that limit their ability to perform walking exercise (including ataxia, peripheral or sensory neuropathy, unstable bone lesion, severe arthritis, pathological lower limb fractures within 6 months, lower limb amputation).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
bone health | baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: C. Ellen Lee, PhD, PT, Principal Investigator — University of Manitoba; Y.K. James Lau, MD, PhD, Principal Investigator — CancerCare Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Lee CE, Leslie WD, Lau YK. A pilot study of exercise in men with prostate cancer receiving androgen deprivation therapy. BMC Cancer. 2012 Mar 21;12:103. doi: 10.1186/1471-2407-12-103. PMID 22436542